CLINICAL TRIAL: NCT05805709
Title: Caring for OutPatiEnts After Acute Kidney Injury (COPE-AKI) Trial
Brief Title: A Patient-centered Trial of a Process-of-care Intervention in Hospitalized AKI Patients: the COPE-AKI Trial
Acronym: COPE-AKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kaleab Abebe, PhD, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY21080024; 1U01DK130010 (NIH); 1U01DK129989 (NIH); 1U01DK129980 (NIH); 1U01DK129984 (NIH)
Record Dates: First submitted 2023-02-23; First posted 2023-04-10 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; process of care; acute renal failure; kidney failure; kidney damage; pragmatic; nurse navigator; pharmacist
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency | interventions — Pharmacists; Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: This is a randomized, pragmatic, parallel-arm kidney trial conducted to find out if an "enhanced care" team approach can improve a patient's outcomes after hospitalization with acute kidney injury (AKI). Participants (N=2145) will be allocated 1:1 to the intervention or usual care using a web-based system to maintain allocation concealment using stratified randomization with randomly permuted blocks. Randomization will be stratified by clinical site.
Who Masked: Outcomes Assessor
Masking Description: Participants and the clinical care teams (nurse navigator, pharmacist, and study physician) will not be masked due to unblinded nature of the intervention. Research coordinators who carry out screening, enrollment, and study visits at baseline, 3, 6 and 12 months will be masked from participant group assignment. Similarly, study visits performed by research coordinator at baseline (enrollment), 3 months and 12 months will be masked. Similarly, assessment of study endpoints will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Process of Care Intervention (Experimental): A multimodal process-of-care intervention that includes 1) study physician oversight and follow up care recommendations at the time of hospital discharge; 2) involvement of a nurse navigator to provide kidney-disease related education, coordinate care, and assess symptoms; and 3) pharmacist-led medication reconciliation and review.
  Interventions: Other: Study Physician/Advance Practice Provider; Other: Nurse Navigator; Other: Pharmacist; Other: Patient Education
- Usual Care (Active Comparator): After receiving the same written information about kidney disease, nephrotoxins to be avoided and importance/need for follow up with a physician as individuals randomized to the multimodal intervention arm, participants randomized to the control arm will receive usual care as specified by their treating providers and will not be followed by nurse navigator, pharmacist, or the study team. The only subsequent study-related activities will be the follow-up study visits for ascertainment of endpoints with the research coordinator.
  Interventions: Other: Patient Education

INTERVENTIONS:
Other: Study Physician/Advance Practice Provider — The nephrologist and/or nephrology-associated advanced practice provider (APP) at each site will lead the intervention team for the duration of the study. The study physicians will fulfil two main roles: (a) Provide supervision to the rest of the study team and (b) conduct a discharge assessment to triage and make recommendations for follow-up care.
  Arms: Multimodal Process of Care Intervention
Other: Nurse Navigator — The nurse navigator will be the primary contact for the participants assigned to the intervention group for the study. The navigator will obtain contact information, information about the patient's usual care providers and pharmacy, review medications, show the participant how to use the home blood pressure machine and scales and arrange for follow-up visits. The role of the nurse navigator will be to monitor the participant's medical condition; facilitate scheduling of needed medical follow-up including both routine (pre-scheduled) and ad hoc (urgent or emergency); enhance adherence with prescribed medical care and follow-up appointments; and serve as a resource to the patient to answer questions about their AKI-related management, facilitate medical and associated care and provide enhanced psychosocial support.
  Arms: Multimodal Process of Care Intervention
Other: Pharmacist — The pharmacist will complete the medication reconciliation and medication regimen review per the predetermined checklist, via telemedicine if agreeable to the patient. The goal of the patient/caregiver-pharmacist interaction is to cover the following: avoidance of nephrotoxins when possible and appropriate, appropriate dosing of renally cleared drugs, review for drug-drug interactions, monitoring appropriate use of chronic medications, medication adherence, monitor for adverse drug reactions, evaluation of non-prescription medication use, medication/disease education and social support.
  Arms: Multimodal Process of Care Intervention
Other: Patient Education — Written information about kidney disease, nephrotoxins to be avoided and importance/need for follow up with a physician will be provided.

SUMMARY:
The COPE-AKI study is a randomized, pragmatic, parallel-arm trial comparing a multimodal intervention to usual care on hospital-free days through 90 days of study follow up. The primary study hypothesis is that patients randomized to the intervention will have increased odds of more hospital-free days through 90 days (primary clinical) compared to those randomized to usual care. Key secondary hypotheses will investigate the impact of the intervention on rates of major adverse kidney events, rates of recurrent AKI, and changes in patient-reported outcomes. Participants (N=2145) will be allocated 1:1 to the intervention or usual care using a web-based system to maintain allocation concealment using stratified randomization with randomly permuted blocks. Randomization will be stratified by clinical site.

DETAILED DESCRIPTION:
The primary study hypotheses for the COPE-AKI study are: compared to usual care, patients randomized to a multimodal intervention will have increased odds of more hospital-free days through 90 days (primary) and lower rates of major adverse kidney events (MAKE) at 180 days, lower rates of recurrent AKI at 180 days, and greater improvements in patient-reported outcomes over 90 days (secondary).

The primary outcome is hospital-free days through 90 days of follow up, defined as 90 minus the number of calendar days in the hospital as either an inpatient or on observation status, based on the determination made by the corresponding hospital. Key secondary outcomes include: rates of MAKE (measured at 90, 180, and 365 days), rates of recurrent AKI (90, 180, and 365 days), and 4 patient-report outcomes: global health related quality of life, AKI-specific health related quality of life, provider interactions, and social support (30, 90, 180, 365 days).

A multimodal process-of-care intervention that includes 1) study physician oversight and follow up care recommendations at the time of hospital discharge; 2) involvement of a nurse navigator to provide kidney-disease related education, coordinate care, and assess symptoms; and 3) pharmacist-led medication reconciliation and review. Participants in the usual care arm will be provided information about their kidney disease, nephrotoxins to be avoided, and the importance of follow up with a physician will be emphasized.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Kidney Disease Improving Global Outcomes (KDIGO) Stage 2/3 AKI with evidence of persistent AKI (defined as meeting Stage 2+ AKI for 2 consecutive days with serum creatinine concentration measurements >12 hours apart)

Exclusion Criteria:

1. AKI due to primary glomerulonephritis, renal vasculitis, or thrombotic microangiopathy
2. Diagnosis of end-stage kidney disease (ESKD) at the time of admission, defined as:

   1. Baseline estimated glomerular filtration rate (eGFR) <15 mL/min/1.73m2
   2. Previous kidney transplant recipient
   3. On chronic dialysis
3. Acute urinary obstruction with rapid kidney function improvement following relief of obstruction
4. Index hospitalization involving nephrectomy
5. Index hospitalization involving solid organ transplant or stem cell/bone marrow transplant
6. Continued dialysis dependence at time of discharge
7. Previous (within 6 months) or new referral to a nephrologist for care specifically for:

   1. Previous or new diagnosis of glomerulonephritis
   2. Primary electrolyte imbalance disorders unrelated to AKI (e.g., syndrome of inappropriate antidiuretic hormone secretion, Bartter syndrome)
   3. Active treatment for acute interstitial nephritis
8. Non-kidney end-organ failure:

   1. Class IV congestive heart failure
   2. Decompensated cirrhosis with Model For End-Stage Liver Disease (MELD) > 30 or those with a diagnosis of hepatorenal syndrome by the clinical teams
   3. End-stage pulmonary disease (advanced stage chronic obstructive pulmonary disease, interstitial lung disease, cystic fibrosis, pulmonary hypertension)
9. Metastatic malignancy or malignancy requiring active treatment (chemotherapy, immunotherapy), such as multiple myeloma
10. Primary goal of care is palliation: life expectancy <6 months
11. Pregnancy
12. Vulnerable populations

    1. Persons incarcerated
    2. Persons institutionalized
13. Inability to provide informed consent

    a. Impaired cognition as demonstrated by the Brief Confusion Assessment Method (bCAM)
14. Concurrent enrollment in a separate greater than minimal risk interventional trial
15. Inability to participate in either in-person or remote visits

    a. Inability to participate as determined by the research team at time of discharge based on disposition (vs uniform decision across site about exclusion based on SNF)
16. Discharge to long-term acute care facility or other hospital-based location

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2145 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2027-03-05 (Estimated)

PRIMARY OUTCOMES:
Hospital-Free Days (HFDs) through day 90 | 90 days
  Hospital-free days through day 90 defined as 90 minus the number of calendar days in the hospital as either an inpatient or on observation status.

SECONDARY OUTCOMES:
Rate of Major Adverse Kidney Events (MAKE) at 180 days | 180 days
  MAKE-180 composite outcome of death, dialysis and assessment of kidney function defined as:
  * death within 180 days of index hospital discharge;
  * need for dialysis at 180 days after index hospital discharge; or
  * serum creatinine >2x baseline at 180 days after index hospital discharge
Recurrent Acute Kidney Injury (AKI) Hospitalization at 180 days | 180 days
  Episodes of recurrent AKI during subsequent all-cause hospitalizations will be adjudicated based on hospitalization data, defining recurrent episodes of AKI based on an increase in serum creatinine of >50% relative to the lowest-known value preceding or including the rehospitalization.
Change from baseline in Global Health-Related Quality of Life (HR-QoL) at 180 days. | 180 days
  HR-QOL will be assessed with the 10-item Patient-Reported Outcomes Measurement Information System (PROMIS) HRQoL measure. The PROMIS Global Health measures assess an individual's physical, mental, and social health. The measures are generic, rather than disease-specific, and often use an "In General" item context as it is intended to globally reflect individuals' assessment of their health. The adult PROMIS Global Health measure produces two scores: Physical Health and Mental Health, which are rescaled into a standardized score (T-score) with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. A higher T-score represents more of the concept being measured. Thus, a person who has T-scores of 60 for the Global Physical Health or Global Mental Health scales is one standard deviation better (more healthy) than the general population.
Change from baseline in AKI-Specific Health-Related Quality of Life (HR-QoL) at 180 days. | 180 days
  AKI-Specific HR-QOL will be assessed with the 6-item Chronic Kidney Disease Quality of Life (CKD-QoL) measure. The CKD-QoL comprehensively represents CKD-specific quality of life and yields a single summary impact score. Norm-based scoring is used (linearly transformed to have a mean of 50 and an SD of 10) in which a higher score indicates worse QOL impact.
Change from baseline in Interactions with Providers at 180 days. | 180 days
  Provider interactions will be assessed with the 5-item Perceived Efficacy in Patient-Physician Interactions (PEPPI) and 8-item Client Satisfaction Questionnaire (CSQ-8) measures. The PEPPI provides a summary score ranging for 5 to 25 (25 = sighted patient self-efficacy). The CSQ-8 is a structured survey used to assess level of satisfaction with care. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with different descriptors for each response point. Total scores range from 8 to 32, with higher scores indicating greater satisfaction.
Change from baseline in Social Support at 180 days. | 180 days
  Social support will be assessed with the 4-item PROMIS Emotional Support and 4-item PROMIS Instrumental Support short forms. The Emotional Support and Instrumental Support measures each produce a summary score, which are rescaled into a standardized score (T-score) with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. A higher T-score represents more of the concept being measured. Thus, a person who has a T-score of 60 is one standard deviation better (more healthy) than the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Kaleab Abebe, PhD, Principal Investigator — Univerisity of Pittsburgh; Linda Fried, MD, Principal Investigator — University of Pittsburgh; Paul Palevsky, MD, Principal Investigator — University of Pittsburgh; Sandy Kane-Gill, PharmD, Principal Investigator — University of Pittsburgh
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Yale University, New Haven, Connecticut
  - Cleveland Clinic Weston Hospital, Weston, Florida
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - MetroHealth, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nashville VA Medical Center, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the University of Pittsburgh Data Coordinating Center (DCC). This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by clinical sites and by the DCC research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived at the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data collected for this study will be analyzed and stored at the University of Pittsburgh Scientific & Data Research Center (SDRC). Six months after publication of the primary manuscript or 18 months after study completion, whichever occurs first, the de-identified, archived data will be transmitted to and stored at the NIDDK Central Repository, for use by other researchers including those outside of the study. Permission to transmit data to the NIDDK Central Repository will be included in the informed consent.